CLINICAL TRIAL: NCT00265759
Title: A Randomized Phase III Trial Comparing 16 to 18 Weeks of Neoadjuvant Exemestane (25 mg Daily), Letrozole (2.5 mg), or Anastrozole (1 mg) in Postmenopausal Women With Clinical Stage II and III Estrogen Receptor Positive Breast Cancer
Brief Title: Exemestane, Letrozole, or Anastrozole in Treating Postmenopausal Women Who Are Undergoing Surgery for Stage II or Stage III Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACOSOG-Z1031; ACOSOG-Z1031; CDR0000456382 (Registry Identifier: NCI Physician Data Query); NCT00698971 (obsolete NCT alias)
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; estrogen receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; exemestane; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Experimental): Patients receive oral exemestane once daily for up to 16-18 weeks.
  Interventions: Drug: exemestane; Procedure: Therapeutic Conventional Surgery
- Arm II (Experimental): Patients receive oral letrozole once daily for up to 16-18 weeks.
  Interventions: Drug: letrozole; Procedure: Therapeutic Conventional Surgery
- Arm III (Experimental): Patients receive oral anastrozole once daily for up to 16-18 weeks.
  Interventions: Drug: anastrozole; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: anastrozole — Given PO
  Arms: Arm III
Drug: exemestane — Given PO
  Arms: Arm I
Drug: letrozole — Given PO
  Arms: Arm II
Procedure: Therapeutic Conventional Surgery — Undergo partial or radical mastectomy or lumpectomy with or without lymph node dissection

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using exemestane, letrozole, or anastrozole, may fight breast cancer by lowering the amount of estrogen the body makes. Giving exemestane, letrozole, or anastrozole before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. It is not yet known whether exemestane, letrozole, or anastrozole is more effective in treating breast cancer.

PURPOSE: This randomized phase III trial is studying exemestane, letrozole, and anastrozole to compare how well they work in treating postmenopausal women who are undergoing surgery for stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether anastrozole, exemestane, or letrozole administered for 16 to 18 weeks as neoadjuvant endocrine treatment for postmenopausal patients with stage II or stage III estrogen receptor (ER)-positive breast cancer should be chosen as the aromatase inhibitor arm of a future study that will compare neoadjuvant aromatase inhibitor (AI) treatment with neoadjuvant chemotherapy. (Cohort A)
* To determine whether patients who have a high Ki-67 value (> 10%) after 2 weeks of neoadjuvant AI treatment experience a higher than expected pathological response rate to neoadjuvant chemotherapy (20%) than would be typically observed for postmenopausal patients with unselected ER+ rich tumors (estimated to be 5%), indicating that an early assessment of proliferation is a useful approach to the identification of a chemotherapy sensitive subgroup of ER+ tumors. (Cohort B [patients enrolled after the 375th patient])

Secondary

* Compare the neoadjuvant treatment regimens relative to the rates of improvement in surgical outcome for patients considered marginal for Breast Conservation Surgery prior to therapy. (Cohort A)
* Compare the neoadjuvant treatment regimens relative to the rates of improvement in surgical outcome for patients designated as candidates for Mastectomy prior to therapy. (Cohort A)
* Compare the relative safety of the neoadjuvant treatment regimens in terms of reported adverse events. (Cohort A)
* To compare the tumor pathologic size between the neoadjuvant treatment regimens, to compare the rates of pathological complete response. (Cohort A)
* To compare the tumor pathologic size between the neoadjuvant treatment regimens, to compare the rates of down-staging to stage I. (Cohort A)
* Compare the incidence of metastatic lymph node involvement on the three arms of the study in patients who have a lymph node dissection at the end of neoadjuvant treatment. (Cohort A)
* Compare the neoadjuvant treatment regimens relative to clinical response rate. (Cohort B)
* Compare the neoadjuvant treatment regimens relative to progression-free survival. (Cohort A and B)
* Compare the neoadjuvant treatment regimens relative to overall survival. (Cohort A and B)

OUTLINE: This is a multicenter study comprising cohort A (phase III study) and cohort B (phase II study). Once cohort A accrual is met (375 patients), subsequent patients are enrolled to cohort B. Patients in both cohorts are stratified according to T stage (T2 vs T3 vs T4), and randomized to 1 of 3 aromatase inhibition (AI) treatment arms.

* Arm I: Patients receive oral exemestane once daily for 16-18 weeks.
* Arm II: Patients receive oral letrozole once daily for 16-18 weeks.
* Arm III: Patients receive oral anastrozole once daily for 16-18 weeks. Patients in cohort B undergo breast biopsy after 2-4 weeks of AI treatment for analysis of Ki-67 levels. Patients with Ki-67 level ≤ 10% continue AI treatment. Patients with Ki-67 level > 10% (high) are given the option to switch to neoadjuvant chemotherapy or undergo immediate breast surgery.

After completion of AI therapy, all patients undergo partial or radical mastectomy or lumpectomy with or without lymph node dissection.

After surgery, patients are followed up periodically for 10 years.

PROJECTED ACCRUAL: A total of 610 patients (375 for cohort A and 235 for cohort B) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

  * T2-T4c, any N, M0 disease
* Clinically staged, as documented by the treating physician, as 1 of the following:

  * T4a-c disease for which modified radical mastectomy with negative margins is the goal
  * T2 or T3 disease for which conversion from needing mastectomy to breast conservation is the goal
  * T2 disease for which lumpectomy at first attempt is the goal
* Primary tumor must be palpable and measure > 2 cm by tape, ruler, or caliper measurements in at least one dimension
* Must agree to undergo mastectomy or lumpectomy after neoadjuvant aromatase inhibitor therapy
* No inflammatory breast cancer, defined as clinically significant erythema of the breast and/or documented dermal lymphatic invasion (not direct skin invasion by tumor or peau d'orange without erythema)
* No distant metastasis (M1)

  * Isolated ipsilateral supraclavicular node involvement allowed
* No diagnosis that was established by incisional biopsy
* Must have estrogen receptor (ER) positive tumor with an Allred score of 6, 7 or 8

  * Patients with > 66.66% (two-thirds) of cells staining positive and have a minimum Allred score of 6 are eligible

PATIENT CHARACTERISTICS:

* ECOG/Zubrod performance status of ≤ 2
* Female
* Patient must be postmenopausal, verified by 1 of the following:

  * Bilateral surgical oophorectomy
  * No spontaneous menses ≥ 1 year
  * No menses for < 1 year with FSH and estradiol levels in postmenopausal range
* No other malignancies within the past 5 years, except for successfully treated cervical carcinoma in situ; lobular carcinoma in situ of the breast; contralateral ductal carcinoma in situ that was treated with mastectomy or lumpectomy with radiotherapy (without tamoxifen); or non-melanoma skin cancer with no evidence of recurrence

  * Must have undergone potentially curative therapy for all prior malignancies AND deemed to be at low risk for recurrence, according to the treating physician

PRIOR CONCURRENT THERAPY:

* No prior treatment for invasive breast cancer, including radiotherapy, endocrine therapy, chemotherapy, or investigational agents
* No prior sentinel lymph node biopsy (cohort B only)
* At least 1 week since prior agents with estrogenic or putatively estrogenic properties, including herbal preparations
* At least 1 week since prior hormone replacement therapy of any type, megestrol acetate, or raloxifene
* No concurrent enrollment in another neoadjuvant clinical trial for treatment of the existing breast cancer
* No other concurrent anti-neoplastic therapy, including chemotherapy or radiotherapy
* No concurrent agents or herbal products that alter ER function

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2019-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Ellis, MD, PhD, FRCP, Study Chair — Washington University Siteman Cancer Center
Locations (3):
- United States (3):
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas

REFERENCES:
- [Result] Ellis MJ, Suman VJ, Hoog J, Lin L, Snider J, Prat A, Parker JS, Luo J, DeSchryver K, Allred DC, Esserman LJ, Unzeitig GW, Margenthaler J, Babiera GV, Marcom PK, Guenther JM, Watson MA, Leitch M, Hunt K, Olson JA. Randomized phase II neoadjuvant comparison between letrozole, anastrozole, and exemestane for postmenopausal women with estrogen receptor-rich stage 2 to 3 breast cancer: clinical and biomarker outcomes and predictive value of the baseline PAM50-based intrinsic subtype--ACOSOG Z1031. J Clin Oncol. 2011 Jun 10;29(17):2342-9. doi: 10.1200/JCO.2010.31.6950. Epub 2011 May 9. PMID 21555689
- [Result] Ellis MJ, Suman VJ, Hoog J, Goncalves R, Sanati S, Creighton CJ, DeSchryver K, Crouch E, Brink A, Watson M, Luo J, Tao Y, Barnes M, Dowsett M, Budd GT, Winer E, Silverman P, Esserman L, Carey L, Ma CX, Unzeitig G, Pluard T, Whitworth P, Babiera G, Guenther JM, Dayao Z, Ota D, Leitch M, Olson JA Jr, Allred DC, Hunt K. Ki67 Proliferation Index as a Tool for Chemotherapy Decisions During and After Neoadjuvant Aromatase Inhibitor Treatment of Breast Cancer: Results From the American College of Surgeons Oncology Group Z1031 Trial (Alliance). J Clin Oncol. 2017 Apr 1;35(10):1061-1069. doi: 10.1200/JCO.2016.69.4406. Epub 2017 Jan 3. PMID 28045625
- [Derived] Punturi NB, Seker S, Devarakonda V, Mazumder A, Kalra R, Chen CH, Li S, Primeau T, Ellis MJ, Kavuri SM, Haricharan S. Mismatch repair deficiency predicts response to HER2 blockade in HER2-negative breast cancer. Nat Commun. 2021 May 19;12(1):2940. doi: 10.1038/s41467-021-23271-0. PMID 34011995

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Z1031A enrolled postmenopausal women with stage II/III ER+ (Allred 6 to 8) breast cancer (BC) whose treatment was randomized to neoadjuvant AI therapy with anastrozole, exemestane or letrozole. For Z1031B the protocol was amended to include a tumor Ki67 determination after 2-4 weeks of AI.
Groups:
- Cohort A Arm I: Exemestane: Patients receive oral exemestane 25 mg once daily for up to 16-18 weeks prior to partial or radical mastectomy or lumpectomy with or without lymph node dissection.
- Cohort A Arm II: Letrozole: Patients receive oral letrozole 2.5 mg once daily for up to 16-18 weeks prior to partial or radical mastectomy or lumpectomy with or without lymph node dissection.
- Cohort A Arm III: Anastrozole: Patients receive oral anastrozole 1 mg once daily for up to 16-18 weeks prior to partial or radical mastectomy or lumpectomy with or without lymph node dissection.
- Cohort B: Patients undergo a core breast biopsy for Ki67 determination after 2 weeks of neoadjuvant aromatase inhibitor (AI) therapy. If the Ki67 was ≤10% the patient continued AI therapy for another 12-14 weeks and then proceeded to surgery. Women whose two-week Ki67 level was > 10% were offered either a NCCN approved neoadjuvant chemotherapy regimen or surgery at the discretion of providers/patients. If the biopsy core contained insufficient tumor to perform the Ki67 assay patients could elect to be re-biopsied at 4 weeks or continue on AI therapy. If severe treatment-related toxicity was reported or the patient refused further AI therapy, surgery was recommended.
Period: Overall Study
Arm/Group | Cohort A Arm I: Exemestane | Cohort A Arm II: Letrozole | Cohort A Arm III: Anastrozole | Cohort B
Started | 124 | 128 | 125 | 245
Completed | 124 | 127 | 123 | 236
Not Completed | 0 | 1 | 2 | 9
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 2
Not completed — Cancel | 0 | 0 | 0 | 3
Not completed — Ineligible | 0 | 0 | 0 | 1
Not completed — Bilateral disease | 0 | 0 | 0 | 2
Not completed — Discontinued due to intolerability | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort B Arm I: Week 2 Ki67 <=10%: Patients undergo a core breast biopsy for Ki67 determination after 2 weeks of neoadjuvant aromatase inhibitor (AI) therapy. If the Ki67 was ≤10% the patient continued AI therapy for another 12-14 weeks and then proceeded to surgery. If severe treatment-related toxicity was reported or the patient refused further AI therapy, surgery was recommended.
- Cohort B Arm II: Week 2 Ki67 >10%: Patients undergo a core breast biopsy for Ki67 determination after 2 weeks of neoadjuvant aromatase inhibitor (AI) therapy. Women whose two-week Ki67 level was > 10% were offered either a NCCN approved neoadjuvant chemotherapy regimen or surgery at the discretion of providers/patients. If severe treatment-related toxicity was reported or the patient refused further AI therapy, surgery was recommended.
- Cohort B Arm III: Week 2 Ki67 No Invasive Disease Present: Patients undergo a core breast biopsy for Ki67 determination after 2 weeks of neoadjuvant aromatase inhibitor (AI) therapy. If the biopsy core contained insufficient tumor to perform the Ki67 assay patients could elect to be re-biopsied at 4 weeks or continue on AI therapy. If severe treatment-related toxicity was reported or the patient refused further AI therapy, surgery was recommended.
- Total: Total of all reporting groups
Arm/Group | Cohort A Arm I: Exemestane | Cohort A Arm II: Letrozole | Cohort A Arm III: Anastrozole | Cohort B Arm I: Week 2 Ki67 <=10% | Cohort B Arm II: Week 2 Ki67 >10% | Cohort B Arm III: Week 2 Ki67 No Invasive Disease Present | Total
Number analyzed (Participants) | 124 | 127 | 123 | 165 | 49 | 22 | 610
Age, Continuous [Median (Full Range); unit: years] | 69 [43 to 90] | 65 [49 to 90] | 65 [51 to 87] | 65 [49 to 86] | 60 [47 to 76] | 66 [53 to 84] | 65 [43 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 127 | 123 | 165 | 49 | 22 | 610
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 124 | 127 | 123 | 165 | 49 | 22 | 610

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response (Complete or Partial Response) Rate (Cohort A)
Description: The clinical response rate (percentage) of a given treatment is defined as 100 times the number of eligible patients randomized to that treatment whose disease meets the WHO criteria for complete or partial response prior to surgery divided by the total number of eligible patients randomized to that treatment. For each treatment arm, a 95% binomial confidence interval will be constructed for the true clinical response rate. Complete Response (CR): The disappearance of all known disease based on a comparison between the measurements at baseline and the Week 16 visit. Partial Response (PR): A 50% or greater decrease in the product of the bi-dimensional measurements of the lesion (total tumor size) based on a comparison between the measurements at baseline and the Week 16 visit. In addition there can be no appearance of new lesions or progression of any lesion.
Time Frame: Up to 18 weeks
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort A Arm I: Exemestane | Cohort A Arm II: Letrozole | Cohort A Arm III: Anastrozole
Number analyzed (Participants) | 124 | 127 | 123
percentage of patients | 62.9 [53.8 to 71.4] | 74.8 [66.3 to 82.1] | 69.1 [60.1 to 77.1]

2. Primary Outcome: Anti-tumor Effect in Terms of Pathologic CR (pCR) Rate to Neoadjuvant Chemotherapy (Cohort B)
Description: The primary aim is to assess the anti-tumor effect in terms of pathologic CR rates of neo-adjuvant chemotherapy in patients with T2-T4c, any N, M0 breast cancer (by clinical staging) who are endocrine therapy resistant (that is, their Ki-67 level is >10 after 2-4 week of neo-adjuvant endocrine therapy alone). The pCR rate (percentage) for neo-adjuvant chemotherapy is defined as 100 times the number of eligible patients with no histologic evidence of invasive tumor cells in the surgical breast specimen and the axillary or sentinel lymph nodes divided by the total number of eligible patients who received neo-adjuvant chemotherapy.
Time Frame: Up to 18 weeks
Population: The Overall Number of Participants Analyzed is a subset of the number of patients in Cohort B Arm II: Week 2 Ki67 >10% who switched to neoadjuvant chemotherapy. The remaining number of patients in this arm were not included in this analysis due to decision to either continue with AI therapy or undergo surgery directly.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Cohort B Arm II: Week 2 Ki67 > 10%: Patients who after 2 weeks of neoadjuvant aromatase inhibitor (AI) therapy had a tumor Ki67 level of greater than 10% and switched to neoadjuvant chemotherapy.
Arm/Group | Cohort B Arm II: Week 2 Ki67 > 10%
Number analyzed (Participants) | 35
percentage of patients | 5.7 [0.7 to 19.1]

3. Secondary Outcome: Toxicity (Cohort A)
Description: Incidence of the most common grade 3+ toxicities reported to be probably, possibly, or definitely related to treatment as assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 (Cohort A) At each treatment evaluation, the type, severity, and attribution of each adverse event reported will be assessed using the NCI-CTCAE definitions. For each treatment, the percentage of patients who developed a severe (grade 3+) toxicity considered possibly, probably or definitively related to treatment will be determined.
Time Frame: Up to 30 days after drug therapy
Measure: Number; unit: percentage of patients
Arm/Group | Cohort A Arm I: Exemestane | Cohort A Arm II: Letrozole | Cohort A Arm III: Anastrozole
Number analyzed (Participants) | 124 | 127 | 123
percentage of patients
  Fatigue | 2 | 2 | 3
  Hot flashes/flushes | 2 | 4 | 2
  Joint pain | 2 | 3 | 2

4. Secondary Outcome: Disease-free Survival (DFS) (Cohort A and B)
Description: Disease-free survival (DFS) is the time from surgery to the first of the following events: local, regional or distant recurrence, second primary disease, contralateral invasive breast cancer, or death due to any cause. The 5 year DFS rate and 95% confidence interval will be calculated.
Time Frame: 5 years
Population: Patients that received treatment and were eligible for analysis were included. Arms are combined across cohorts for survival analysis, as defined in the protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort A: Patients receive oral letrozole, anastrozole, or exemestane once daily for up to 16-18 weeks prior to partial or radical mastectomy or lumpectomy with or without lymph node dissection
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 334 | 192
percentage of participants | 84.5 [80.5 to 88.7] | 87.4 [82.6 to 92.5]

5. Secondary Outcome: Rate of Improved Surgical Outcome for Patients Considered Marginal for Breast Conservation Surgery Prior to Therapy (Cohort A)
Description: The rate (percentage) of improved surgical outcome for patients considered marginal for breast conservation surgery prior to therapy for Cohort A is reported below for each treatment arm. Breast conservation surgery (not mastectomy) as the most extensive surgery performed for a patient is considered an improvement in surgical outcome.
Time Frame: At time of surgery up to 18 weeks
Population: Overall Number of Participants Analyzed only includes patients considered marginal for breast conservation surgery prior to therapy.
Measure: Number (95% Confidence Interval); unit: percentage of improved surgical outcome
Arm/Group | Cohort A Arm I: Exemestane | Cohort A Arm II: Letrozole | Cohort A Arm III: Anastrozole
Number analyzed (Participants) | 61 | 62 | 66
percentage of improved surgical outcome | 85.2 [73.3 to 92.6] | 77.4 [64.7 to 86.7] | 86.4 [75.2 to 93.2]

6. Secondary Outcome: Rate of Downstaging to Stage I Determined by Sentinel Node Evaluation (Cohort A)
Description: The rate downstaging to Stage I of a given treatment is defined as 100 times the number of eligible patients randomized to that treatment whose surgically findings are such that the maximum dimension of the invasive lesion contained in their surgical specimen is at most 2 cm and their lymph nodes are negative (by Hematoxylin & Eosin Staining) divided by the total number of eligible patients randomized to that treatment. For each neo-adjuvant endocrine treatment pair, a 95% binomial confidence interval will be constructed for the true difference in the rate of downstaging to Stage I between these 2 treatments.
Time Frame: At time of surgery up to 18 weeks
Population: Outcome Measure Data Not Collected.
Arm/Group | Cohort A Arm I: Exemestane | Cohort A Arm II: Letrozole | Cohort A Arm III: Anastrozole
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Rate of Lymph Node Involvement (LNI) (Cohort A)
Description: For those patients who undergo a sentinel lymph node dissection or an axillary lymph node dissection (at least 6 nodes examined with Hematoxylin & Eosin Staining), the LNI rate (percentage) is defined as 100 times the proportion of eligible patients randomized to that treatment with at least one positive node. For each neo-adjuvant endocrine treatment, a 95% binomial confidence interval will be constructed for its true LNI rate.
Time Frame: At time of surgery up to 18 weeks
Population: Overall Number of Participants Analyzed include only patients who were evaluated for the number of positive nodes and not evaluated before or during AI therapy.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort A Arm I: Exemestane | Cohort A Arm II: Letrozole | Cohort A Arm III: Anastrozole
Number analyzed (Participants) | 107 | 112 | 111
percentage of patients | 41.1 [31.8 to 51.1] | 48.2 [38.7 to 57.8] | 44.1 [34.8 to 53.9]

8. Secondary Outcome: The Pathologic Complete Response (pCR) Rate (Cohort A)
Description: The pathologic complete response is defined as no histologic evidence of invasive tumor cells in the surgical breast specimen and axillary or sentinel lymph nodes. The pathologic complete response rate (percentage) of a given treatment is defined as 100 times the number of eligible patients randomized to that treatment whose surgical specimen is such that there is no histologic evidence of invasive tumor cells in the surgical breast specimen and axillary or sentinel lymph nodes divided by the total number of eligible patients randomized to that treatment. For each neo-adjuvant endocrine treatment pair, a 95% binomial confidence interval will be constructed for the true difference in the pCR between these 2 treatments.
Time Frame: At time of surgery up to 18 weeks
Population: Overall Number of Participants Analyzed only includes patients who had surgery performed after completion of AI therapy.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort A Arm I: Exemestane | Cohort A Arm II: Letrozole | Cohort A Arm III: Anastrozole
Number analyzed (Participants) | 115 | 120 | 117
percentage of patients | 1.7 [0.3 to 6.8] | 0.0 [0.0 to 3.9] | 0.0 [0.0 to 4.0]

9. Secondary Outcome: Clinical Response Rate (Cohort B)
Description: The clinical response rate is defined as 100 times the number of eligible patients whose disease meets the WHO criteria for complete or partial response prior to surgery divided by the total number of eligible patients. A 90% binomial confidence interval will be constructed for the true clinical response rate.
Time Frame: Up to 18 weeks
Population: Outcome Measure Data Not Collected.
Arm/Group | Cohort B
Number analyzed (Participants) | 0

10. Secondary Outcome: Rate of Improved Surgical Outcome for Patients Designated as Candidates for Mastectomy Prior to Therapy (Cohort A)
Description: Rate (percentage) of Improved surgical outcome for patients designated as candidates for mastectomy prior to therapy (Cohort A). Breast conservation surgery (not mastectomy) as the most extensive surgery performed for a patient is considered an improvement in surgical outcome.
Time Frame: At time of surgery up to 18 weeks
Population: Overall Number of Participants Analyzed only includes patients considered candidates for mastectomy prior to therapy.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort A Arm I: Exemestane | Cohort A Arm II: Letrozole | Cohort A Arm III: Anastrozole
Number analyzed (Participants) | 52 | 57 | 50
percentage of patients | 48.1 [34.0 to 62.4] | 42.1 [29.1 to 55.9] | 60.0 [49.2 to 77.1]

11. Secondary Outcome: Percentage of Participants With Overall Survival (Cohort A and B)
Description: Overall survival (OS) will be measured from the date of randomization until the date of death. The distribution of overall survival times will be estimated using the Kaplan-Meier method. The 5 year OS rate and 95% confidence interval will be calculated.
Time Frame: 5 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 334 | 192
percentage of participants | 88.1 [84.6 to 91.7] | 88.6 [84.1 to 93.3]

ADVERSE EVENTS:
Time Frame: Adverse events are assessed at the following time points: at W4, W8, W12, Within 1 week of W16, W16, and 30 days post drug therapy; Up to 10 years.
Description: This study will collect adverse events using the Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE v.3.0). Note that effective April 1, 2011, CTCAE Version 4 has been used for expedited reporting via AdEERS. All graded adverse events are reported.
Arm/Group | Cohort A Arm I: Exemestane | Cohort A Arm II: Letrozole | Cohort A Arm III: Anastrozole | Cohort B
Serious Adverse Events (participants affected / at risk) | 9/157 | 14/157 | 12/155 | 5/144
Other Adverse Events (participants affected / at risk) | 146/157 | 146/157 | 140/155 | 123/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Arm I: Exemestane (N=157) | Cohort A Arm II: Letrozole (N=157) | Cohort A Arm III: Anastrozole (N=155) | Cohort B (N=144)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (3) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dental prosthesis user (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (3) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (3) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 10 (11) | 5 (7) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General symptom (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Small intestine infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Small intestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (7) | 3 (5) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (4) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 5 (5) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 3 (4) | 1 (2) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 8 (8) | 3 (5) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A Arm I: Exemestane (N=157) | Cohort A Arm II: Letrozole (N=157) | Cohort A Arm III: Anastrozole (N=155) | Cohort B (N=144)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 5 (9) | 0 (0)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (5) | 1 (1) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 3 (6) | 0 (0)
Cardiac pain (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 5 (8) | 2 (6)
Ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (6) | 3 (13) | 1 (2) | 0 (0)
Hearing test abnormal (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (6) | 0 (0) | 0 (0)
Endocrine disorder (Endocrine disorders) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Cataract (Eye disorders) | 1 (5) | 1 (5) | 1 (2) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (3) | 2 (3) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 1 (1) | 2 (2) | 3 (5) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flashing vision (Eye disorders) | 0 (0) | 1 (5) | 2 (3) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 2 (6) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (4) | 4 (10) | 0 (0) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (4) | 2 (2)
Anal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 14 (23) | 14 (24) | 12 (22) | 13 (19)
Dental prosthesis user (Gastrointestinal disorders) | 1 (1) | 1 (4) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 24 (40) | 11 (16) | 11 (16) | 5 (9)
Dry mouth (Gastrointestinal disorders) | 3 (5) | 2 (6) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (4) | 1 (6)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 2 (4) | 0 (0) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (4) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 5 (5) | 1 (1) | 5 (9) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 39 (59) | 41 (70) | 36 (57) | 23 (44)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary gland disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 12 (15) | 11 (21) | 12 (16) | 3 (3)
Chest pain (General disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Chills (General disorders) | 2 (3) | 1 (3) | 1 (2) | 0 (0)
Edema limbs (General disorders) | 10 (20) | 8 (20) | 12 (19) | 6 (9)
Fatigue (General disorders) | 94 (280) | 88 (230) | 87 (230) | 76 (221)
Fever (General disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Flu-like symptoms (General disorders) | 1 (1) | 1 (4) | 1 (1) | 0 (0)
General symptom (General disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Injection site reaction (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders) | 2 (3) | 2 (3) | 2 (5) | 1 (1)
Pain (General disorders) | 6 (8) | 7 (13) | 11 (13) | 6 (8)
Autoimmune disorder (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune system disorder (Immune system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (2) | 1 (1)
Bronchitis (Infections and infestations) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gingival infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Infection (Infections and infestations) | 4 (4) | 3 (3) | 3 (3) | 1 (1)
Lip infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 1 (1) | 5 (6) | 4 (4)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (2) | 2 (2) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 5 (5) | 4 (4) | 2 (2) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 3 (5) | 2 (4) | 3 (3) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 4 (4) | 0 (0)
Intraoperative musculoskeletal injury - Extremity-upper (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraoperative venous injury - Vein-jugular (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 3 (4) | 2 (3) | 2 (2) | 4 (4)
Wound dehiscence (Injury, poisoning and procedural complications) | 5 (6) | 1 (1) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 3 (5) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Coagulopathy (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 3 (9) | 1 (1)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 2 (6) | 1 (1)
Leukocyte count decreased (Investigations) | 0 (0) | 1 (1) | 2 (6) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (3) | 1 (1)
Serum cholesterol increased (Investigations) | 0 (0) | 1 (1) | 1 (5) | 1 (1)
Weight gain (Investigations) | 3 (3) | 0 (0) | 2 (3) | 1 (1)
Weight loss (Investigations) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 6 (9) | 8 (16) | 5 (9) | 3 (4)
Blood glucose increased (Metabolism and nutrition disorders) | 5 (8) | 4 (6) | 4 (6) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 75 (218) | 75 (205) | 77 (189) | 57 (152)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (8) | 2 (5) | 1 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 39 (84) | 36 (97) | 40 (99) | 27 (63)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 1 (3) | 2 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Developmental disturbance (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibrosis (Musculoskeletal and connective tissue disorders) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Joint disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (5) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 25 (40) | 19 (51) | 28 (50) | 13 (34)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 (5) | 5 (5) | 2 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 38 (73) | 41 (83) | 41 (93) | 27 (58)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (5) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (6) | 7 (11) | 5 (9) | 3 (10)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper extremity dysfunction (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (5)
Dizziness (Nervous system disorders) | 20 (28) | 17 (32) | 11 (19) | 7 (9)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 3 (5) | 1 (3)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Glossopharyngeal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 29 (59) | 37 (75) | 37 (62) | 20 (38)
Memory impairment (Nervous system disorders) | 3 (4) | 7 (12) | 2 (7) | 0 (0)
Mini mental status examination abnormal (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 2 (3) | 2 (6) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 14 (30) | 9 (16) | 11 (16) | 8 (13)
Sinus pain (Nervous system disorders) | 2 (3) | 2 (2) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 21 (38) | 19 (34) | 29 (51) | 11 (23)
Anxiety (Psychiatric disorders) | 40 (77) | 42 (82) | 48 (96) | 29 (64)
Confusion (Psychiatric disorders) | 1 (2) | 1 (1) | 3 (3) | 1 (1)
Depression (Psychiatric disorders) | 32 (73) | 29 (64) | 32 (63) | 21 (37)
Euphoria (Psychiatric disorders) | 2 (3) | 5 (12) | 6 (11) | 0 (0)
Insomnia (Psychiatric disorders) | 18 (34) | 12 (21) | 12 (22) | 15 (40)
Bladder pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cystitis (Renal and urinary disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 4 (9) | 4 (4) | 1 (6) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 3 (6) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Breast hypoplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 12 (19) | 13 (21) | 17 (27) | 14 (30)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (5) | 1 (1)
Reproductive tract disorder (Reproductive system and breast disorders) | 1 (2) | 1 (2) | 1 (1) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 2 (5) | 3 (4) | 3 (7) | 1 (5)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 4 (16) | 5 (13) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 14 (33) | 8 (18) | 6 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 (45) | 24 (52) | 20 (52) | 13 (34)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngoscopy abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5) | 2 (2) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 1 (4) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (11) | 4 (8) | 5 (15) | 5 (13)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (3) | 2 (5) | 2 (2) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (5) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (11) | 9 (19) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 5 (6) | 4 (5) | 3 (3) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 7 (10) | 3 (4) | 7 (10) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 7 (10) | 4 (4) | 4 (7) | 3 (8)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (5) | 1 (1)
Hematoma (Vascular disorders) | 3 (3) | 4 (4) | 2 (2) | 1 (1)
Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hot flashes (Vascular disorders) | 77 (241) | 103 (330) | 86 (296) | 82 (277)
Hypertension (Vascular disorders) | 6 (11) | 10 (24) | 14 (33) | 7 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes